CLINICAL TRIAL: NCT05124223
Title: Analysis of Cardiac Damage Post Infection With SARS-CoV-2 and Post Vaccination Against COVID-19
Status: Completed | Type: Observational
Sponsor: Sebastian Kelle (Other)
Responsible Party: Sponsor-Investigator, Sebastian Kelle, Head of cardiovascular MRI, German Heart Institute
Organization: German Heart Institute (Other)
Other Study IDs: EA2/020/21
Record Dates: First submitted 2021-11-16; First posted 2021-11-17 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Myocarditis Acute
Keywords: COVID-19; COVID-19-Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-COVID-19: From May 2020 to May 2021, we retrospectively examined 104 clinical cardiac magnetic resonance (CMR) examinations performed in patients with suspected cardiac involvement post COVID-19. The mean time from first positive PCR to CMR was 112 +- 76 days. During their COVID-19 disease, 21% of patients required hospitalization, 17% supplemental oxygen and 7% mechanical ventilation.
  Interventions: Diagnostic Test: Cardiac MRI
- Post-COVID-19-Vaccination: Between May 2021 and August 2021, we examined 27 patients with suspected cardiac disease after COVID-19 vaccination.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Cardiac MRI was performed as clinically indicated to assess cardiac pathology.

SUMMARY:
From May 2020 to May 2021, the investigators retrospectively evaluated clinical cardiac magnetic resonance (CMR) examinations performed in patients with suspected cardiac involvement post COVID-19. Between May 2021 and August 2021, the investigators evaluated patients with suspected cardiac disease after COVID-19 vaccination.

DETAILED DESCRIPTION:
Hospital database for patients that underwent a clinical CMR examination between May 2020 and May 2021 for suspected cardiac pathology post COVID-19 were analyzed. For comparison, CMR examinations from January until August 2021 were searched for suspected cardiac pathology post COVID-19 vaccination. The study complies with the declaration of Helsinki and was approved by the ethics committee of the Charité-Universitätsmedizin Berlin (EA2/020/21).

CMR Imaging All scans were performed for clinical indications on either a Philips Ingenia 3.0 T scanner or a Philips Ambition 1.5 T scanner according to recent recommendations for CMR in patients post COVID-19. Protocols were adjusted to the clinical scenario but generally included standard CINE imaging, T2 STIR edema imaging, basal and medial short axis T2 mapping (T2-GraSE) and pre- and post-contrast T1 mapping (MOLLI), and Late-Enhancement-Imaging (mDIXON). Vasodilator stress with Regadenosone or Adenosine was performed in patients with clinically suspected myocardial ischemia. The Adenosine dose was 0.140 µg/kg/min, with an increase to 0.210 µg/kg/min in case of insufficient response. The Regadenosone dose was 200µg irrespective of weight, followed by Theophyllin reversal as needed (max. 200mg). The contrast agent was 0.1 mmol/kg Gadobutrol (Gadovist®, Bayer AG, Leverkusen, Germany).

CMR image analysis Image post-processing and measurements were performed according to recent recommendations using dedicated CMR post-processing software (IntelliSpace Portal V11.1, Philips, Best, The Netherlands). The diagnosis of 'probable myocarditis' was based on the updated Lake Louise Criteria requiring findings of myocardial damage (LGE) and edema (T2 STIR or T2 mapping) in a non-ischemic pattern (intramyocardial or subepicardial). Evidence of edema without myocardial damage was considered 'possible myocarditis' whereas myocardial damage without edema was considered 'subsided myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac MRI for suspected cardiac Involvement after COVID-19 or COVID-19-vaccination

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical all-comers with suspected cardiac Involvement after COVID-19 or COVID-19-vaccination
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Acute Myocarditis | January 2020 to August 2021
  Number of patients with CMR diagnosis of suspected acute myocarditis

SECONDARY OUTCOMES:
Subsided Myocarditis | January 2020 to August 2021
  Number of patients with CMR diagnosis of suspected subsided myocarditis

CONTACTS AND LOCATIONS:
Locations (1):
- German Heart Center Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No